CLINICAL TRIAL: NCT00429312
Title: A Phase I/II, Open-Label Study of JX-594 (Thymidine Kinase-deleted Vaccinia Virus Plus GM-CSF) Administered by Intratumoral Injection in Patients With Unresectable Stage 3 or Stage 4 Malignant Melanoma
Brief Title: A Study of Recombinant Vaccinia Virus to Treat Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX594-IT-MEL005
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2010-03

CONDITIONS: Melanoma
Keywords: Melanoma; Oncolytic virus; Pexa-Vec
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Intratumoral injection(s) of Recombinant Vaccinia GM-CSF, JX-594
  Interventions: Biological: JX-594

INTERVENTIONS:
Biological: JX-594 — Thymidine kinase-deleted vaccinia virus plus GM-CSF
  Other Names: JX594

SUMMARY:
The purpose of this research study is to find out whether JX-594 (Pexa-Vec) is safe and effective for treating surgically unresectable malignant melanoma.

DETAILED DESCRIPTION:
Cancer of the skin is the most common of all cancers, probably accounting for more than 50% of all cancers. Melanoma accounts for about 4% of skin cancer cases but causes a large majority of skin cancer deaths. The American Cancer Society estimates that about 62,190 new melanomas will be diagnosed in the United States during 2006.

DTIC is the only chemotherapy drug approved by the FDA for the treatment of metastatic melanoma. The reported response rates are 5-20% without any evidence of prolonged survival in randomized clinical trials versus best supportive care. The median overall survival for melanoma patients treated with DTIC alone is approximately 8 months; PFS and TTP following treatment with DTIC is approximately 7 weeks, and the objective response rate for DTIC alone (CR+PR) is less than 10% (Millward, 2004). Other chemotherapy agents including cisplatin and carboplatin, BCNU, vindesine, paclitaxel, docetaxel, and vinorelbine have also been tested but none have improved upon the very modest activity of DTIC.

Melanoma may be the optimal target for JX-594 immunotherapy because of the relatively high rate of accessible disease for injection, the positive response of melanoma seen with IL-2 immunotherapy, and the lack of effective, tolerable therapy for patient with metastatic melanoma. Furthermore, it is speculated that JX-594 replication targets the EGFR pathway, which is highly expressed in melanocytes.

Results from an initial Phase I/II study suggest that intratumoral injection of JX-594 is safe and effective in treating both injected and distant disease in patients with surgically incurable metastatic melanoma. Response of both injected tumors (in 5 of 7 patients) and response of at least one non-injected tumor (in 4 of 7 patients) was demonstrated, including two patients who achieved a partial response (6 + months) and a complete response (4 + months) to JX-594 treatment. Particularly noteworthy is that efficacy and gene expression occurred despite pre-treatment vaccination (and, therefore, pre-existing anti-vaccinia immunity) in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, Stage 3 or Stage 4 malignant melanoma
* At least one tumor mass measurable by CT/MRI and/or physical examination that can be injected by direct visualization or by ultrasound-guidance
* Anticipated survival of at least 16 weeks
* Cancer is not surgically resectable for cure
* KPS score of ≥ 70 (refer to APPENDIX E: KARNOFSKY PERFORMANCE STATUS (KPS))
* Age ≥18 years
* Men and women of reproductive potential must be willing to follow accepted birth control methods during treatment and for 3 months after the last treatment with JX-594
* The ability to understand and willingness to sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent form
* Able to comply with study procedures and follow-up examinations
* Adequate liver function: Total bilirubin ≤ 2.0 x ULN; AST, ALT ≤ 2.0 x ULN
* Adequate bone marrow function: WBC > 3,500 cells/mm3 and < 50,000 cells/mm3; ANC > 1,500 cells/mm3; Hemoglobin > 10 g/dL; Platelet count > 125,000 plts/mm3
* Acceptable coagulation status: INR < (ULN + 10%)
* Acceptable kidney function: Serum creatinine < 2.0 mg/dL

Exclusion Criteria:

* Target tumor(s) adherent to and/or invading a major vascular structure (e.g. carotid artery)
* Pregnant or nursing an infant
* Known infection with HIV
* Systemic corticosteroid or other immunosuppressive medication use within 4 weeks of first treatment with JX-594
* Clinically significant active infection or uncontrolled medical condition (e.g. pulmonary, neurological, cardiovascular, gastrointestinal, genitourinary) considered high risk for investigational new drug treatment Significant immunodeficiency due to underlying illness and/or medication (e.g. systemic corticosteroids)
* History of eczema that at some stage has required systemic therapy
* Clinically significant and/or rapidly accumulating ascites, peri-cardial and/or pleural effusions (e.g. requiring drainage for symptom control)
* Severe or unstable cardiac disease which includes, but is not limited to, any of the following within 6 months prior to screening: myocardial infarct, unstable angina, congestive heart failure, myocarditis, arrhythmias diagnosed and requiring medication, or any clinically-significant change in cardiac status
* Treatment of the target tumor(s) with radiotherapy, chemotherapy, surgery, or an investigational drug within 4 weeks of screening (6 weeks in case of mitomycin C or nitrosoureas)
* Experienced a severe reaction or side-effect as a result of a previous smallpox vaccination
* Inability or unwillingness to give informed consent or comply with the procedures required in this protocol
* Patients with household contacts who are pregnant or nursing an infant, children < 5 years old, have history of eczema that at some stage has required systemic therapy, or have a significant immunodeficiency due to underlying illness (e.g. HIV) and/or medication (e.g. systemic corticosteroids) will be excluded unless alternate living arrangements can be made during the patient's active dosing period and for three weeks following the last dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Response rate for injected tumor(s) | Initial response assessment at 6 weeks

SECONDARY OUTCOMES:
Safety, as determined by incidence of treatment-related adverse events, serious adverse events (SAEs), and clinically-significant changes from baseline in routine laboratory parameters | Safety evaluation throughout study period
Best overall response for entire disease burden (RECIST criteria) | Initial response assessment after six weeks
Progression-free survival (PFS) | Follow-up every three weeks until new therapy or disease progression
Response rate of non-injected tumor(s) | Initial response assessment at six weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Burke, M.D., Principal Investigator — Billings Clinic; David H Kirn, M.D., Study Director — Jennerex Biotherapeutics
Locations (3):
- United States (3):
  - UCLA, Los Angeles, California
  - Billings Clinic, Billings, Montana
  - Cancer Center of the Carolinas, Greenville, South Carolina

REFERENCES:
- [Background] Mastrangelo MJ, Maguire HC Jr, Eisenlohr LC, Laughlin CE, Monken CE, McCue PA, Kovatich AJ, Lattime EC. Intratumoral recombinant GM-CSF-encoding virus as gene therapy in patients with cutaneous melanoma. Cancer Gene Ther. 1999 Sep-Oct;6(5):409-22. doi: 10.1038/sj.cgt.7700066. PMID 10505851